CLINICAL TRIAL: NCT07407855
Title: Comparative Evaluation of Giomer-Based Composite Restorations in Class V Carious Lesions in Diabetic Versus Non-Diabetic Patients Using Modified USPHS Criteria: An 18-Month Non-Randomized Clinical Trial
Brief Title: Clinical Performance of Giomer-Based Composite Restorations in Class V Carious Lesions in Diabetic and Non-Diabetic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Wael Maher, Lecturer Assistant, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU-FD-CD-4-1-3-2025
Record Dates: First submitted 2026-01-25; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic Patients (Experimental): Controlled diabetic patients with Class V carious lesions restored using Giomer-based composite resin
  Interventions: Device: Giomer-based composite restoration
- Non-Diabetic Patients (Active Comparator): Non-diabetic patients with Class V carious lesions restored using the same Giomer-based composite and adhesive protocol.
  Interventions: Device: Giomer-based composite restoration

INTERVENTIONS:
Device: Giomer-based composite restoration — Giomer-based composite restoration (Beautifil® II LS, SHOFU, USA) using universal adhesive (BeautiBond® Xtreme, SHOFU, USA).

SUMMARY:
Diabetes mellitus is associated with structural and biochemical alterations in dentin that may negatively affect the clinical performance and longevity of adhesive dental restorations, particularly in cervical carious lesions. Giomer-based composite resins, containing pre-reacted glass ionomer fillers, release fluoride and other beneficial ions that may enhance remineralization and reduce the risk of secondary caries.

This prospective, parallel-group, non-randomized clinical trial aims to evaluate the clinical performance of Giomer-based composite restorations in Class V carious lesions in controlled diabetic and non-diabetic patients. Restorations will be assessed using Modified USPHS criteria at baseline, 6, 12, and 18 months, with retention as the primary outcome and marginal adaptation, secondary caries, marginal discoloration, and post-operative sensitivity as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Class V carious lesions (ICDAS scores 3 or 4).
* Controlled diabetic patients diagnosed with diabetes mellitus (for diabetic group).
* Non-diabetic patients with no systemic diseases (for control group).
* Teeth indicated for Class V composite restoration.

Exclusion Criteria:

* Uncontrolled diabetes mellitus.
* Patients with other systemic diseases affecting oral health.
* Teeth with pulpal involvement or requiring endodontic treatment.
* Patients with parafunctional habits. Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Restoration Retention Score Assessed Using Modified USPHS Criteria | Baseline, 6 months, 12 months, and 18 months
  Retention of Class V Giomer-based composite restorations will be evaluated using Modified United States Public Health Service (USPHS) criteria. Each restoration will be assigned an ordinal score (Alpha, Bravo, Charlie) based on the presence or loss of restoration. Data will be reported as distribution of USPHS scores and frequency of restoration loss over time.

SECONDARY OUTCOMES:
Marginal Adaptation Score Assessed Using Modified USPHS Criteria | Baseline, 6 months, 12 months, and 18 months
  Marginal integrity between tooth and restoration will be evaluated using Modified USPHS criteria. Each restoration will receive an ordinal score (Alpha, Bravo, Charlie) at each follow-up visit.
Secondary Caries Score Assessed Using Modified USPHS Criteria | Baseline, 6 months, 12 months, 18 months
  Presence of recurrent caries adjacent to the restoration will be assessed using Modified USPHS criteria and recorded as ordinal categorical scores (Alpha, Bravo, Charlie).
Marginal Discoloration Score Assessed Using Modified USPHS Criteria | Baseline, 6 months, 12 months, 18 months
  Discoloration at the tooth-restoration margin will be evaluated using Modified USPHS criteria and recorded as ordinal categorical scores.
Post-Operative Sensitivity Score Assessed Using Modified USPHS Criteria | Baseline, 6 months, 12 months, 18 months
  Tooth sensitivity associated with restored teeth will be clinically evaluated and scored using Modified USPHS criteria ordinal scores.

IPD SHARING:
Plan to Share IPD: Undecided